CLINICAL TRIAL: NCT03839212
Title: Preventing Cardiometabolic Disease in HIV-Infected Latino Men Through a Culturally-Tailored Health Promotion Intervention
Brief Title: The Happy Older Latinos Are Active (HOLA) Health Promotion Study in HIV-Infected Latino Men
Acronym: HOLAHIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Daniel Enrique Jimenez, Associate Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20181032; U54MD002266 (NIH)
Record Dates: First submitted 2019-02-08; First posted 2019-02-15 (Actual); Results first posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-07

CONDITIONS: Human Immunodeficiency Virus; Cardiometabolic Risk
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Happy Older Latinos are Active (HOLA) (Experimental): A 16-week multi-component, health promotion intervention
  Interventions: Behavioral: HOLA Component 1; Behavioral: HOLA Component 2; Behavioral: HOLA Component 3; Behavioral: HOLA Component 4

INTERVENTIONS:
Behavioral: HOLA Component 1 — At week 1 and week 8 participants will meet individually with Community Health Worker (CHW) for 30 minutes for a manualized social and physical activation session.
Behavioral: HOLA Component 2 — A CHW led 45 minute (10 minutes of stretching and warm up, followed by 30 minutes of walking with a 5 minute cool down) group walk session of six participants at a time done 3 times a week that utilized interval training that slowly gradually increases in intensity.
Behavioral: HOLA Component 3 — A CHW led pleasant event discussion, asking each participant to identify a pleasant event. This task is done in conjunction with the cool down of HOLA 2.
Behavioral: HOLA Component 4 — One booster walking session twice a month for three months post intervention for reinforcement.

SUMMARY:
The purpose of this study is to examine the feasibility of an intervention to prevent chronic diseases like diabetes, high blood pressure, and obesity in midlife and older Latino adults living with HIV. The investigators expect that the participant will be in this study for seven months. Participants will be interviewed and asked to take part in walking groups.

ELIGIBILITY:
Inclusion Criteria:

* are Latino (self-identified);
* are age 50+ years;
* are male;
* are HIV infected but are virologically suppressed (viral load <200 copies/mL);
* volunteer informed consent;
* have medical clearance by a physician;
* expect to stay in Miami for the next 6 months; and
* have documented risk of cardiometabolic disease.

Exclusion Criteria:

* diabetes diagnosis;
* at baseline meet criteria for current major depressive disorder or generalized anxiety disorder;
* meet criteria for current alcohol or other substance abuse disorders;
* have a lifetime history of bipolar disorder or other psychotic disorder;
* have a diagnosis of any neurodegenerative disorder or dementia (Parkinson's disease, Alzheimer's, vascular, frontotemporal dementia, etc.) or significant cognitive impairment as indicated by a Mini Mental Status Exam score <24;
* have contraindications to physical activity outlined in the American College of Sports Medicine standards;
* have high suicide risk i.e., intent or plan to attempt suicide in the near future (a response of "yes" to questions 3, 4, and/or 5 on the Paykel Questionnaire);
* are unable to complete 10 m walk test;
* currently residing in a nursing or group home;
* have a terminal physical illness expected to result in the death within one year;
* have an acute or severe medical illness that precludes them from safely participating in a health promotion intervention.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2020-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Jimenez, Ph.D., Principal Investigator — University of Miami
Locations (1):
- Jackson Memorial Mental Health Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jimenez DE, Weinstein ER, Batsis J. You gotta walk the walk to talk the talk: protocol for a feasibility study of the Happy Older Latino Adults (HOLA) health promotion intervention for older HIV-positive Latino men. Pilot Feasibility Stud. 2023 Feb 28;9(1):32. doi: 10.1186/s40814-023-01262-w. PMID 36855194

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Happy Older Latinos Are Active (HOLA)
Started | 18
Completed | 14
Not Completed | 4
Not completed — COVID-19 related suspension of research activities. | 4

BASELINE CHARACTERISTICS:
Arm/Group | Happy Older Latinos Are Active (HOLA)
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Eligible Participants Refusing to Participate.
Description: Number of eligible participants refusing to participate.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Happy Older Latinos Are Active (HOLA)
Number analyzed (Participants) | 18
Participants | 0

2. Primary Outcome: Retention Rate
Description: Retention rate will be reported as the number of participants completing the post-intervention assessment.
Time Frame: Up to 3 months post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Happy Older Latinos Are Active (HOLA)
Number analyzed (Participants) | 18
Participants | 14

3. Primary Outcome: Acceptability of Intervention
Description: As measured by the total number of sessions attended by the participants as a whole.
Time Frame: Up to week 16
Measure: Number; unit: sessions
Arm/Group | Happy Older Latinos Are Active (HOLA)
Number analyzed (Participants) | 18
sessions | 111

4. Secondary Outcome: Change in Cardiometabolic Risk as Measured by Waist Circumference
Description: As measured by the number of inches around the participant's waist. A waist circumference of 102 centimetres (40 inches) or more in men is associated with health problems such as type 2 diabetes, heart disease and high blood pressure.
Time Frame: Baseline, 7 months post intervention
Reporting Status: Not Posted

5. Secondary Outcome: Change in Psychosocial Functioning as Measured by Depression Severity Scale
Description: As measured by a 20-item Center for Epidemiologic Studies Depression (CES-D) scale. The possible range of scores are 0 to 60 with the higher scores indicating the presence of more symptomatology.
Time Frame: Baseline, Month 4, Month 7
Reporting Status: Not Posted

6. Secondary Outcome: Change in Health-related Quality of Life as Measured by the Short Form Health Survey (SF-12)
Description: The SF-12v2 is a measure of health related quality of life and provides 2 scores 1) Mental Component Summary Score (MCS) and 2) Physical Component Summary Score (PCS). MCS scores range from 0 to 100, higher scores indicate better mental health related quality of life.
Time Frame: Baseline, Month 4, Month 7
Reporting Status: Not Posted

7. Secondary Outcome: Change in Psychosocial Functioning as Measured by the Patient Health Questionnaire (PHQ-9)
Description: severity of depression will be measured by the 9-item PHQ-9. Scores range from 0 to 27. With scores of 1-4 indicating minimal depression and scores of 20-27 indicating severe depression.
Time Frame: Baseline, Month 4, Month 7
Reporting Status: Not Posted

8. Secondary Outcome: Change in Psychosocial Functioning as Measured by the Severity of Anxiety Using the Generalized Anxiety Disorder Scale
Description: The 7-item Generalized Anxiety Disorder (GAD-7) scale will be used to measure the severity of anxiety. The scores range from 0 to 21 with scores of 0 to 5 indicating mild anxiety and scores of 15-21 indicating severe anxiety.
Time Frame: Baseline, Month 4, Month 7
Reporting Status: Not Posted

9. Secondary Outcome: Change in Psychosocial Functioning as Measured by the Severity of Anxiety Using the Perceived Stress Scale
Description: The 14 item Healthy Families Program Perceived Stress Scale will be used to measure the severity of anxiety. PSS scores can range from 0 to 40 with higher scores indicated higher perception of stress.
Time Frame: Baseline, Month 4, Month 7
Reporting Status: Not Posted

10. Secondary Outcome: Change in Psychosocial Functioning as Measured by the Social Support Received
Description: The 12 item Multidimensional Scale of Perceived Social support. After calculating the mean score across the categories a mean scale support score from 1 to 2.9 would indicate low support, whereas a mean score of 5.1 to 7 would indicate high support.
Time Frame: Baseline, Month 4, Month 7
Reporting Status: Not Posted

11. Secondary Outcome: Change in Lipid Profile as Measured by Total Cholesterol, HDL-C, LDL-C, Triglycerides
Description: A total cholesterol value of less than 200 mg/dL (5.18 mmol/L) is desirable and 240 mg/dL (6.22 mmol/L) or higher is high. Average HDL-C level is 40-50 mg/dL (1.0-1.3 mmol/L) for men. Low HDL-C level, increased risk, is less than 40 mg/dL (1.0 mmol/L). Optimal LDL-C levels are less than 100 mg/d while high levels are 160-189 mg/dL (4.15-4.90 mmol/L). Desirable triglyceride levels are less than 150 mg/dL (1.70 mmol/L) while high levels are considered 200-499 mg/dL (2.3-5.6 mmol/L).
Time Frame: Baseline, Month 4, Month 7
Reporting Status: Not Posted

12. Secondary Outcome: Change in Hypertension as Measured by Systolic and Diastolic Blood Pressure.
Description: Normal systolic and diastolic pressure is less than 120 mmHg and 80mmHg, respectively. High systolic and diastolic pressure is 140 mmHg or higher and 90 mmHg or higher, respectively.
Time Frame: Baseline, Month 4, Month 7
Reporting Status: Not Posted

13. Secondary Outcome: Change in Glucose as Measured by Glycated Hemoglobin (Hba1c)
Description: The normal range for the hemoglobin A1c level is between 4% and 5.6%. Hemoglobin A1c levels between 5.7% and 6.4% mean a higher chance of getting diabetes. Levels of 6.5% or higher mean diabetes.
Time Frame: Baseline, Month 4, Month 7
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Happy Older Latinos Are Active (HOLA)
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

LIMITATIONS AND CAVEATS:
All clinical research activities at the University of Miami were suspended due to the Coronavirus Disease of 2019 (COVID-19) pandemic. As a result, data collection and participant retention were impacted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/12/NCT03839212/Prot_SAP_001.pdf
  • Informed Consent Form (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/12/NCT03839212/ICF_000.pdf